CLINICAL TRIAL: NCT06416566
Title: The Efficacy of Low-Dose Enoxaparin in Psoriasis
Brief Title: Low-Dose Enoxaparin in Psoriasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Norhan Anees, Principal Investigator, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Enoxaparin in psoriasis
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enoxaparin (Experimental): will receive subcutaneous enoxaparin
  Interventions: Drug: Subcutaneous Enoxaparin

INTERVENTIONS:
Drug: Subcutaneous Enoxaparin — Selected patients will receive subcutaneous low dose enoxaparin once a week for 6 weeks.The level of serum heparinase enzyme will be measured before and after treatment

SUMMARY:
Rationale:

* Psoriasis is a chronic immune-mediated inflammatory skin disorder where T cells play a fundamental role in its pathogenesis.
* Low molecular weight heparin has been reported to exert immunomodulatory effect at small doses through inhibition of T cells heparinase enzyme.
* Low molecular weight heparin may have promising results for treatment of psoriasis.

Research question:

* Can low molecular weight heparin be used safely for treatment of psoriasis with good outcome?
* Is enoxaparin inhibitory effect on T cell heparinase enzyme responsible for its beneficial effect?

Hypothesis:

* Low molecular weight heparin can achieve good results when used at small doses for treatment of psoriasis.
* Heparin can exert immunomodulatory effect in psoriasis through inhibition of T cell heparinase enzyme.

AIM OF WORK

-The aim of this work is to assess the possible clinical efficacy and safety of low-dose enoxaparin in the treatment of psoriasis and to detect if inhibition of heparinase enzyme might account for its beneficial therapeutic effect.

Objectives:

* To evaluate safety and efficacy of low molecular weight heparin at small dose for treatment of psoriasis.
* Contribute to the ongoing efforts to optimize psoriasis management and improve the lives of individuals affected by this chronic condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with plaque psoriasis, who met the following criteria will be enrolled.

  1. Age 18 and above.
  2. No systemic (oral, parenteral, photobiological) treatment for psoriasis within the last 2 months.
  3. No topical treatment for psoriasis within the last 2 weeks.

Exclusion Criteria:

* 1. Pregnancy or lactation. 2. Hypersensitivity to heparin and heparin derivatives and a history of heparin-induced thrombocytopenia.

  3. History of bleeding diathesis, uncontrolled hypertension, cerebrovascular accident, peptic ulcer, liver disease and/or abnormal liver function tests or abnormal kidney function tests.

  4. History of major surgery within the last 3 months. 5. A family history of bleeding diathesis, or cerebrovascular accident. 6. Concomitant use of oral anticoagulants, acetylsalicylic acid, or other nonsteroidal anti-inflammatory drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Psoriatic Area and Severity Index score | weekly for 6 weeks and at follow up period of 6 weeks
  The studied patients will be clinically evaluated weekly for 6 weeks and at follow up period; biweekly for 6 weeks

IPD SHARING:
Plan to Share IPD: Undecided